CLINICAL TRIAL: NCT03252119
Title: High Flow Oxygen Therapy vs Standard Care in Infants With Viral Bronchiolitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High flow oxygen therapy became available as standard care
Sponsor: Chris Hani Baragwanath Academic Hospital (Other)
Responsible Party: Principal Investigator, Susan Murphy, Specialist Intensivist, Chris Hani Baragwanath Academic Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M170234
Record Dates: First submitted 2017-05-04; First posted 2017-08-17 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Bronchiolitis, Viral
MeSH Terms: conditions — Bronchiolitis, Viral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard therapy group (No Intervention): standard treatment of viral bronchiolitis with low flow oxygen.
- high flow humidified oxygen group (Experimental): treatment of viral bronchiolitis with high flow humidified oxygen therapy.
  Interventions: Device: High flow humidified oxygen therapy

INTERVENTIONS:
Device: High flow humidified oxygen therapy — application of high flow humidified oxygen therapy at 2l/kg/min
  Arms: high flow humidified oxygen group

SUMMARY:
A randomized control trial of 130 infants admitted to the paediatric high care admission ward will be enrolled, and randomized to either "high flow humidified oxygen" or "standard therapy".

DETAILED DESCRIPTION:
A randomized control trial of 130 infants admitted to the paediatric high care admission ward will be enrolled. Infants between 1 month and 2 years of age who fulfill criteria for enrollment shall be considered eligible. Informed consent from parents or legal guardians shall be obtained. Infants shall be randomized to either "standard therapy" or "high flow humidified oxygen". Measurements of heart rate, respiratory rate, work of breathing (Tal score and WCAS), oxygen saturation and oxygen requirements shall be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of viral bronchiolitis
* Not requiring intubation and ventilation
* Admitted to high care unit
* With moderate/severe respiratory distress (Tal score >6)
* Saturations <92% in room air

Exclusion Criteria:

* congenital cardiac disease
* presence of multiorgan failure/multisystemic disease
* previously ventilated
* craniofacial abnormalities
* nasal pathology
* decreased level of consciousness
* Ex-prem <34 weeks
* Possible impending respiratory failure

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Effect of high flow humidified oxygen therapy on work of breathing | during first 5 days post enrollment
  Respiratory rate (n/min)
Effect of high flow humidified oxygen therapy on work of breathing | first 5 days post enrollment
  Use of accessory muscles of respiration (present /not)
Effect of high flow humidified oxygen therapy on blood oxygen saturations | first 5 days post enrollment
  Saturation of oxygen (% saturation) as measured by pulse oximeter
Effect of high flow humidified oxygen therapy on heart rate | first 5 days post enrollment
  Pulse (n/min) measured by ECG monitor

SECONDARY OUTCOMES:
Proportion of patients requiring intubation and ventilation | from time of enrollment to end of hospital stay (up to 6 months)
  number of patients (N) getting intubated
Length of hospital stay | from time of enrollment to end of hospital stay (up to 6 months)
  days (N) spent in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Murphy, FCPaed (SA), Principal Investigator — University of the Witwatersrand, Johannesburg
Locations (1):
- Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No
No plan to share data wit other researchers